CLINICAL TRIAL: NCT05091996
Title: The Application of Manual Techniques in Masticatory Muscles Relaxation as Adjunctive Therapy in the Treatment of Temporomandibular Joint Disorders
Brief Title: The Use of Manual Muscle Relaxation Techniques in the Treatment of Temporomandibular Joint Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Bartosz Trybulec, Principal Investigator, Jagiellonian University
Allocation: Non-Randomized | Model: Parallel | Purpose: Supportive Care
Other Study IDs: 122.6120.129.2016
Record Dates: First submitted 2021-09-28; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Temporomandibular Disorder; Temporomandibular Joint Disorders
Keywords: Temporomandibular disorder; Physiotherapy
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Myofascial Release Therapy

ARMS (2):
- Post-isometric muscle relaxation group (Experimental): The post-isometric relaxation techniques were administered to the mandibular adductors and muscles responsible for lateral movements of the mandible.
  Interventions: Procedure: Post-isometric muscle relaxation technique
- Myofascial release group (Experimental): The myofascial release procedure was performed successively in the area of the anterior parts of the temporal muscles, the superficial parts of the masseter muscles and the sternocleidomastoid muscles.
  Interventions: Procedure: Myofascial release technique

INTERVENTIONS:
Procedure: Post-isometric muscle relaxation technique — 1: Therapist (T) abducted the patients' (P) mandible until the functional barrier. P performed isometric tension of the mandibular adductors with about 20% of the maximum force, balanced by the T. After 10 secs of isometric tension, P relaxed his muscles, and T abducted the mandible to a new functional barrier. During one treatment, the cycle was repeated 3 times, each time starting from the previously obtained barrier.
  2: T performed passive lateral translation of the mandible until the functional barrier. P performed isometric tension with about 20% of maximum force, as to initiate the movement of the mandible towards the resting position. T balanced the force generated by the P. After 10 secs of isometric tension, P relaxed his muscles and T deepened the lateral movement of the mandible until a new functional barrier was reached. During one treatment, the cycle was repeated 3 times, both to the right and left side, each time starting from the previously obtained barrier.
  Arms: Post-isometric muscle relaxation group
Procedure: Myofascial release technique — The myofascial release procedure was performed successively in the area of: the anterior parts of the temporal muscles , the superficial parts of the masseter muscles and the sternocleidomastoid muscles.During one session, the above cycle was repeated six times on both sides separately. The was lying on his back, with his head turned to the side.The therapist was behind the patient's head, using the pad of the first finger placed on the skin in the area of the initial attachment of a worked muscle, he took out the tissue slack, moving the tissues towards the perceptible limitation of mobility (caudal direction).Reaching the tissue barrier, he kept the tension of the sliding structures, shifting them until the physiological tissue barrier.A single application of the myofascial release procedure consisted of one movement moving the soft tissues along the muscle
  Arms: Myofascial release group

SUMMARY:
The aim of the study was to compare the degree of relaxation of the anterior part of the temporal muscles and the masseter muscles achieved with the use of post-isometric relaxation and myofascial release methods in patients requiring prosthetic treatment due to temporomandibular joint disorders (TMD) with a dominant muscular component.

The study included 60 patients, both sexes, aged between 19 and 40. The patients who met the inclusion criteria were alternately assigned to one of the two study groups: I group consisted of the patients received post-isometric relaxation treatment (PIR), II group - patients received myofascial release treatment (MFR). Each group consisted of 30 subjects. The series of ten treatments were performed in both groups. The comparative assessment was carried out based on the data obtained from the physical examination, physiotherapeutic examination of the masticatory system, surface electromyography (sEMG) of anterior temporal and masseter muscles and the data on the intensity of spontaneous masticatory muscle pain assessed using the Visual Analogue Scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* diagnosed functional disorders of the masticatory system with the accompanying excessive tension of the masseter muscles,
* no clinical signs of displacement of the disc with a blockage in the temporomandibular joint,
* spontaneous pain in the masticatory muscles, lasting at least one month before treatment,
* good general health of the patient,
* full dental arches
* written consent to participate in the study

Exclusion Criteria:

* occurrence of a face or head injury during participation in the research project,
* open wounds in the area where the therapy was carried out,
* sudden illness of the patient preventing participation in the study,
* the will to terminate participation in the study

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change From Baseline Electrical Activity of the Anterior Part of the Temporal and Masseter Muscles at 10, and 14 days | Change From Baseline Electrical Activity of the Muscles at 10, and 14 days; Triple measurement: immediately before supportive treatment, after the last of the 10 relaxation treatments and on the 4th day after the end of therapy
  The electrical activity of the anterior part of the temporal and masseter muscles was assessed by surface electromyography (sEMG). The assessment was performed using a two-channel device - NeuroTrac MyoPlus 4 (Verity Medical Ltd.) and surface electrodes (Noraxon inc.). Examination of the same muscles on the right and left sides of the body was performed at the same time. The muscle tone of the anterior part of the temporal muscles was assessed first, followed by the masseter muscles. The parameter describing the degree of electrical activity of the muscle was the mean value of the thirty-second sEMG measurement.
Change From Baseline in Muscle Pain Scores on the Visual Analog Scale at 10, and 14 days | Change From Baseline in Muscle Pain Scores on the Visual Analog Scale at 10, and 14 days; Triple measurement: immediately before supportive treatment, after the last of the 10 relaxation treatments and on the 4th day after the end of therapy
  Assessment of the intensity of spontaneous pain in the masticatory muscles The intensity of spontaneous pain in the masticatory muscles was assessed on the basis of a 10-point visual analogue scale(VAS).This scale included 11 pain grades- from 0 to 10,where 0 was no pain at all, 5 was moderate pain, and 10 was the strongest pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Bartosz Trybulec, PhD, Study Chair — Jagiellonian University Medical College in Cracow

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: starting from the time when summary data are published
Access Criteria: via e-mail on request